CLINICAL TRIAL: NCT03657407
Title: Belladonna and Opium Rectal Suppository Effect on Postoperative Pain and Nausea Following Total Laparoscopic and Robotic-Assisted Hysterectomy
Brief Title: B&O for TLH Post-operative Pain and Nausea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anna Reinert (Other)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor-Investigator, Anna Reinert, Study coordinator, Resident Physician, Mercy Medical Center
Organization: Mercy Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMC 2015-63
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Hysterectomy; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomization to one-time intervention A (medicated suppository) or intervention B (placebo), allocation was sealed in consecutively numbered opaque envelopes generated by biostatistician using blocked randomized technique.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelopes generated by biostatistician used to determine intervention A or B. Drug dictionary entries created within the Pyxis system by the Mercy Medical Center Department of Pharmacy, as "Protocol Drug A" and "Protocol Drug B", recorded in medical record in this way. Identity of "Protocol Drug A" and "Protocol Drug B" revealed by pharmacist at conclusion of data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- B&O (Active Comparator): 29 women randomized to Belladonna & Opium suppository
  Interventions: Drug: Belladonna Opium
- Placebo (Sham Comparator): 27 women randomized to Glycerin suppository
  Interventions: Drug: Glycerin Suppository

INTERVENTIONS:
Drug: Belladonna Opium — Belladonna Opium 16.2-60mg rectal suppository
  Arms: B&O
Drug: Glycerin Suppository — Glycerine rectal suppository
  Arms: Placebo

SUMMARY:
A prospective, single-center, double-blind, randomized, placebo-controlled trial to assess the impact of immediate post-operative placement of a Belladonna and Opium (B&O) rectal suppository on postoperative pain and nausea following laparoscopic and robot-assisted hysterectomy.

DETAILED DESCRIPTION:
This study is a single-center, double-blind, randomized placebo-controlled trial to assess the impact of immediate postoperative Belladonna and Opium rectal suppository use on postoperative pain and nausea following total laparoscopic and robot-assisted hysterectomy. Study took place at Mercy Medical Center, involving both outpatient and inpatient surgical settings. The duration of the trial was 12 months, with 56 patients enrolled during this time period. Patients eligible for trial participation were women between ages 18 and 75 undergoing level I total laparoscopic or robot-assisted hysterectomy with or without bilateral salpingo-oophorectomy, with or without cystoscopy performed post-procedure, with or without lysis of adhesions, and with or without surgical treatment of endometriosis, with no additional surgical procedures being performed (i.e. no lymph node dissection or urogynecologic suspension or sling procedures). Patients were excluded from the study if they had contraindications to the use of B&O suppositories: these contraindications are glaucoma, severe hepatic or renal disease, bronchial asthma, history of narcotic idiosyncracies, respiratory depression, convulsive disorders, acute alcoholism or delirium tremens, or regular use of an anticholinergic medication (twice per week or more frequently). Patients were withdrawn from the study if the original planned surgery was not performed. If the original planned surgery was not performed, a suppository was not placed following surgery. There were no financial incentives offered for trial participation.

Only the patients of clinical investigators from this trial were considered for participation in this study. Clinical investigators posting patients for total laparoscopic or robotic hysterectomy at Mercy Medical Center informed patients of the presence of the clinical trial at the time of surgical posting, using an IRB-approved script. The chart number of patients posted for total laparoscopic or robot-assisted hysterectomy was be forwarded to the co-investigator by the clinic surgical coordinator at the time of surgical posting. The co-investigator reviewed each chart and conducted a telephone interview with each patient prior to surgery to verify trial eligibility and to answer any questions about the trial. Patients were made aware that study participation is voluntary, and that if they chose to not participate, they would receive standard postoperative pain and nausea pharmacologic management. On the day of surgery, a member of the research team met with the patient pre-operatively in a private pre-operative holding area to review and sign a written consent for participation in the trial. This member of the research team was familiar with the study protocol and risks of the pharmacologic intervention under investigation. These steps allowed patients to be fully informed, and ensured patient safety and support during the short interval of the study.

On the day of surgery, patients were randomized to either B&O rectal suppository or to a placebo of glycerin rectal suppository. This study employed a glycerin rectal suppository as a placebo because this over-the-counter medication has limited effects, similar to those of a Belladonna & Opium Supprette, and is similar in size, physical appearance and mechanical properties to a Belladonna & Opium Supprette. A placebo-free comparison group was not used, as this would have changed the study design from a double-blind clinical trial to a single-blind clinical trial, with greater potential for investigator bias to influence study results. Additionally, it is not thought that results for a placebo-free comparison group would substantially differ from those of a glycerin suppository placebo group, and would require a larger study population and greater study resources to achieve findings of similar significance and power. Randomization was performed by a biostatistician, with a sealed envelope created for each patient containing information regarding randomization to either placebo or intervention group. In the operating room, this envelope was opened, and the circulating nurse would draw the indicated medication from the Pyxis system. Drug dictionary entries were created within the Pyxis system by the Mercy Medical Center Department of Pharmacy, so that the Belladonna & Opium Supprette #16A (16.2mg / 60mg), and the glycerin suppository were represented as "Protocol Drug A" and "Protocol Drug B". The patient's electronic medical record reflected that "Protocol Drug A" or "Protocol Drug B" was received by the patient, so that the nurses and physicians caring for the patient postoperatively were blinded as to which suppository the patient received.

A suppository was placed rectally by a member of the surgical team at the conclusion of surgery, prior to departure from the OR and awakening from anesthesia. Post-operative placement was selected to minimize interaction with intraoperative anesthetic and analgesic medications, to maximize peak plasma concentrations and therapeutic efficacy of Belladonna alkaloids and Opium within the immediate postoperative period, and control for variation in procedure length between study participants. The nurses caring for the patient postoperatively were blinded to which suppository the patient did receive, but were made aware that the patient had received a suppository containing either glycerin or one containing belladonna 16.2mg and opium 60mg, equivalent to approximately 6mg of morphine. The nurses were be educated about potential side effects of Belladonna & Opium suppositories, and of potential drug interactions; they were asked to document and to inform the covering provider of the occurrence of any such adverse effects. Patients remaining in the hospital overnight following their surgery underwent a postoperative exam by a resident physician familiar with the study protocol and familiar with potential side effects of the B&O suppository. Standard of care at Mercy Medical Center is for nurses to assess patient's postoperative pain by visual analog scale at regular time intervals. Data regarding patients' visual analog pain scores for the first 12 hours following surgery were extracted from the electronic medical record and analyzed by the research team. PO and IV narcotic use in IV morphine equivalents, PO and IV NSAIDs, and PO and IV antiemetic use were also assessed over the first 12 following surgery, this data was extracted from the electronic medical record and analyzed by the research team. Study surveillance did not extend beyond the duration of the participant's postoperative hospitalization, usually less than 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* between ages 18 and 75,
* undergoing level I total laparoscopic or robot-assisted hysterectomy with or without bilateral salpingo-oophorectomy, cystoscopy, lysis of adhesions, or surgical treatment of endometriosis

Exclusion Criteria:

* contraindications to the use of B&O (i.e. glaucoma, severe hepatic or renal disease, bronchial asthma, history of narcotic idiosyncracies, respiratory depression, convulsive disorders, acute alcoholism or delirium tremens, or regular use of an anticholinergic medication (twice per week or more frequently)
* additional surgical procedures being performed

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Audlin, MD, Principal Investigator — Surgeon
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A cohort of 281 women was assessed for trial eligibility. Patients were excluded from enrollment if the patient could not be reached pre-operatively (n=47), if inclusion criteria were not met (n=67), or if participation was declined (n=106). A cohort of 61 women met criteria for trial enrollment.
Pre-assignment Details: From a cohort of 61 women meeting criteria for trial enrollment, individuals were excluded from study participation and randomization if the study protocol was not executed by the surgical team i.e. study medication was not ordered/administrated (n=5). 56 women underwent randomization/assignment to the study interventions.
Groups:
- Belladonna & Opium: 29 women randomized to Belladonna & Opium suppository
  Belladonna Opium: Belladonna Opium 16.2-60mg rectal suppository
Period: Overall Study
Arm/Group | Belladonna & Opium | Placebo
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belladonna & Opium | Placebo | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (7.9) | 41.8 (6.2) | 43.1 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 56
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Pain-related indication for surgery [Count of Participants; unit: Participants] — Pre-operative diagnosis of pelvic pain, dysmenorrhea, or dyspareunia
  Participants | 18 | 16 | 34
Robotic surgery [Count of Participants; unit: Participants] | 14 | 13 | 27
Laparoscopic surgery [Count of Participants; unit: Participants] | 15 | 14 | 29
Performed by a high-volume surgeon [Count of Participants; unit: Participants] | 19 | 16 | 35
Surgery length [Mean (Standard Deviation); unit: minutes] | 97.7 (49.7) | 96.0 (49.5) | 96.9 (49.2)
Planned admission for 23-hour observation [Count of Participants; unit: Participants] | 8 | 5 | 13
Dexamethasone while under anesthesia [Count of Participants; unit: Participants] | 29 | 26 | 55
Lidocaine while under anesthesia [Count of Participants; unit: Participants] | 27 | 26 | 53
Ketorolac while under anesthesia [Count of Participants; unit: Participants] | 23 | 25 | 48
Zofran while under anesthesia [Count of Participants; unit: Participants] | 21 | 19 | 40
Reglan while under anesthesia [Count of Participants; unit: Participants] | 17 | 16 | 33
Scopolamine patch pre-operatively [Count of Participants; unit: Participants] | 1 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain: VAS
Description: Visual analog pain scale (VAS) (0 to 10, 0 = no pain, 10 = maximum pain), averaged over duration of PACU stay until discharge criteria met
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belladonna & Opium | Placebo
Number analyzed (Participants) | 29 | 27
score on a scale | 4.1 (2.9) | 4.8 (2.1)
Statistical Analysis 1: Comparison: Belladonna & Opium vs Placebo; Null hypothesis that Belladonna & Opium not superior to Placebo; Test type: Superiority; p = 0.17, t-test, 1 sided; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-0.71 to 2.0]

2. Secondary Outcome: Narcotic Use
Description: Cumulative oral and intravenous narcotics received in PACU until PACU discharge criteria met
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalents in mg
Arm/Group | Belladonna & Opium | Placebo
Number analyzed (Participants) | 29 | 27
Oral Morphine Equivalents in mg | 19.3 (14.2) | 21.3 (13.5)
Statistical Analysis 1: Comparison: Belladonna & Opium vs Placebo; Null hypothesis that Belladonna & Opium not superior to Placebo; Test type: Superiority; p = 0.29, t-test, 1 sided; Mean Difference (Final Values) = -2.02, 95% CI 2-sided [-5.4 to 9.5]

3. Secondary Outcome: Time Until Cleared for PACU Discharge
Description: Time elapsed from conclusion of surgery until criteria for PACU discharge met
Time Frame: up to 4 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Belladonna & Opium | Placebo
Number analyzed (Participants) | 29 | 27
minutes | 91.3 (36.7) | 110.6 (51.4)
Statistical Analysis 1: Comparison: Belladonna & Opium vs Placebo; Null hypothesis that Belladonna & Opium not superior to Placebo; Test type: Superiority; p = 0.05, t-test, 1 sided; Median Difference (Final Values) = -19.31, 95% CI 2-sided [-43.1 to 4.5]

4. Secondary Outcome: Number of Participants for Which Anti-emetics Were Received in PACU
Description: Binary assessment of whether anti-emetics received in PACU
Time Frame: up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Belladonna & Opium | Placebo
Number analyzed (Participants) | 29 | 27
Participants | 10 | 11
Statistical Analysis 1: Comparison: Belladonna & Opium vs Placebo; Null hypothesis that Belladonna & Opium not superior to Placebo; Test type: Superiority; p = 0.42, t-test, 1 sided; Mean Difference (Final Values) = 0.85, 95% CI 2-sided [0.42 to 1.7]

ADVERSE EVENTS:
Time Frame: Duration of PACU stay (up to 4 hours)
Arm/Group | Belladonna & Opium | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

LIMITATIONS AND CAVEATS:
Study was limited by low power; sample size at 50% of target by power calculations.

Pre-operative scopolamine patch use was not controlled within study randomization, and varied significantly between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03657407/Prot_SAP_ICF_000.pdf